CLINICAL TRIAL: NCT03611829
Title: An ACT-Based Physician-Delivered Weight Loss Intervention
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The trial was ended prematurely due to low recruitment/enrolment.
Sponsor: McGill University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 405-0316; CIHR PJT-153383 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2018-06-18; First posted 2018-08-02 (Actual); Results first posted 2019-08-14 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2018-12

CONDITIONS: Overweight and Obesity; Eating Behavior
Keywords: emotional eating
MeSH Terms: conditions — Overweight; Obesity; Feeding Behavior; Emotional Eating | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: The present study was a two-arm pilot randomized controlled trial.
Who Masked: Participant
Masking Description: Participants were blind to their condition, but physicians and administrative staff were not blind to participant condition. Physicians were not blind to participant condition because they were responsible for delivering the ACT intervention or standard care. They were thus required to know the participant's condition in order to deliver the adequate treatment. Administrative staff was responsible for providing physicians with this information and organizing study paperwork and thus needed to be aware of participant condition as well.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (Active Comparator): Participants in the standard care condition were provided with diet and exercise counselling and psychoeducation from their physicians over the course of 8 sessions, as was routinely done at the clinic. Standard care did not involve any targeted intervention to reduce emotional eating.
  Interventions: Behavioral: Standard Care
- ACT Intervention (Experimental): In addition to receiving standard care, participants in the ACT condition were taught techniques to reduce their emotional eating. Three overarching skills were taught over the course of the ACT intervention: (1) values clarification and commitment, (2) metacognitive awareness, and (3) distress tolerance. Throughout the sessions, physicians formed if-then plans with the patients to specify how to habitually use the ACT techniques to reduce emotional eating in their everyday lives. At the end of each session, participants were given a one-page homework sheet that asked them to monitor their behavior and their use of the ACT techniques during the week.
  Interventions: Behavioral: ACT Intervention; Behavioral: Standard Care

INTERVENTIONS:
Behavioral: ACT Intervention
  Arms: ACT Intervention
Behavioral: Standard Care

SUMMARY:
The purpose of the present study was to conduct a pilot RCT to test the feasibility of a physician-delivered ACT-based intervention for emotional eaters with overweight/obesity against standard care at a network of weight loss clinics. Participants were randomized to receive either standard care at the clinics or the ACT intervention.

DETAILED DESCRIPTION:
The purpose of the present study was to conduct a pilot RCT to test the feasibility of a physician-delivered ACT-based intervention for emotional eaters with overweight/obesity against standard care at a network of weight loss clinics. Psychology clinical PhD students trained physicians in the delivery of the brief manualized intervention and were available for regular consults. The intervention consisted of eight, 5-10 minute sessions that could be easily incorporated into the physician's current practice. Over the duration of the ACT intervention, physicians met individually with patients to teach them various techniques to address and improve mindfulness, acceptance, and values clarification and commitment, all of which emotional eaters have been found to struggle with (Forman & Butryn, 2014). The proven habit formation technique of if-then planning (Gollwitzer, 1993) was used throughout these sessions in order to train emotional eaters to habitually use ACT techniques and to change the maladaptive habit of eating in response to negative emotions.

ELIGIBILITY:
Inclusion Criteria:

* Only participants considered to be emotional eaters, as assessed by a score of 3.25 or higher on the Dutch Eating Behavior Questionnaire (DEBQ), were recruited for the study (van Strien, Herman, Anschutz, Engels, & de Weerth, 2012).

Exclusion Criteria:

* Not being an emotional eater.
* Participants who did not speak, write, and read in English fluently were excluded from the study, as well as those who were pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2016-05-07 (Actual); Primary Completion 2018-03-07 (Actual); Study Completion 2018-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mallory Frayn, PhD (c), Principal Investigator — McGill University; Kimberly Carrière, PhD Student, Study Director — McGill University; Bärbel Knäuper, PhD, Principal Investigator — McGill University

IPD SHARING:
Plan to Share IPD: Yes
Study data, including the intervention manual, study protocol, statistical analysis plan, and outcomes will be shared with other researchers upon request.
Supporting Information: Study Protocol, SAP
Time Frame: Upon publication of the study results.
Access Criteria: Upon request from other researchers.

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Care: Participants in the standard care condition were provided with diet and exercise counselling and psychoeducation from their physicians over the course of 8 sessions, as was routinely done at the clinic. Standard care did not involve any targeted intervention to reduce emotional eating.
  Standard Care
- ACT Intervention: In addition to receiving standard care, participants in the ACT condition were taught techniques to reduce their emotional eating. Three overarching skills were taught over the course of the ACT intervention: (1) values clarification and commitment, (2) metacognitive awareness, and (3) distress tolerance. Throughout the sessions, physicians formed if-then plans with the patients to specify how to habitually use the ACT techniques to reduce emotional eating in their everyday lives. At the end of each session, participants were given a one-page homework sheet that asked them to monitor their behavior and their use of the ACT techniques during the week.
  ACT Intervention
  Standard Care
Period: Overall Study
Arm/Group | Standard Care | ACT Intervention
Started | 43 | 44
Completed | 21 | 19
Not Completed | 22 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Care | ACT Intervention | Total
Number analyzed (Participants) | 43 | 44 | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.87 (15.18) | 46.94 (14.21) | 46.91 (14.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 31 | 61
  Male | 13 | 13 | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 15 | 24 | 39
Region of Enrollment [Number; unit: participants]
  Canada | 43 | 44 | 87
DEBQ Emotional Eating [Mean (Standard Deviation); unit: units on a scale] — The emotional eating subscale of the Dutch Eating Behavior Questionnaire. Scores range from 1 (never) to 5 (very often). Lower scores reflect lower emotional eating. This subscale score is calculated by taking the mean of all items on the subscale.
  units on a scale | 4.09 (0.53) | 3.96 (0.49) | 4.02 (0.51)
DEBQ External Eating [Mean (Standard Deviation); unit: units on a scale] — The external eating subscale of the Dutch Eating Behavior Questionnaire. Scores range from 1 (never) to 5 (very often). Lower scores reflect lower external eating. This subscale score is calculated by taking the mean of all items on the subscale.
  units on a scale | 3.57 (0.65) | 3.56 (0.56) | 3.56 (0.60)
DEBQ Restraint Eating [Mean (Standard Deviation); unit: units on a scale] — The restraint eating subscale of the Dutch Eating Behavior Questionnaire. Scores range from 1 (never) to 5 (very often). Lower scores reflect lower restraint eating. This subscale score is calculated by taking the mean of all items on the subscale.
  units on a scale | 3.18 (0.64) | 3.17 (0.69) | 3.17 (0.66)
DTS Total Score [Mean (Standard Deviation); unit: units on a scale] — This is the total score of the Distress Tolerance Scale. All items were rated on a 5-point Likert scale from 1 (strongly agree) to 5 (strongly disagree). The score is calculated as the mean of all items. Higher scores reflect higher levels of distress tolerance.
  units on a scale | 2.48 (0.94) | 2.69 (0.84) | 2.59 (0.89)
PHLMS awareness [Mean (Standard Deviation); unit: units on a scale] — This is the awareness subscale of the Philadelphia Mindfulness Scale. All items were rated on a 5-point Likert scale from 1 (never) to 5 (very often). The subscale score is calculated as the sum of all items on the subscale, with the minimum possible score being 10 and the maximum possible score being 50. Higher scores reflect higher levels of awareness.
  units on a scale | 36.03 (6.02) | 36.06 (6.78) | 36.04 (6.38)
PHLMS acceptance [Mean (Standard Deviation); unit: units on a scale] — This is the acceptance subscale of the Philadelphia Mindfulness Scale. All items were rated on a 5-point Likert scale from 1 (never) to 5 (very often). The subscale score is calculated as the sum of all items on the subscale, with the minimum possible score being 10 and the maximum possible score being 50. Higher scores reflect higher levels of acceptance.
  units on a scale | 24.94 (7.79) | 26.00 (7.00) | 25.50 (7.34)
ACT assessment [Mean (Standard Deviation); unit: units on a scale] — This questionnaire was developed for the present study to evaluate participants' real world application of the intervention. Participants were asked to indicate their level of agreement on a 5-point scale (1 = strongly agree and 5 = strongly disagree) to prompts such as "My values motivate me to lose weight" and "I am able to accept negative emotions and don't have to eat when I'm feeling bad". Total score was calculated as the mean of all items. Lower scores indicate better application of the skills learned from the intervention.
  units on a scale | 2.92 (0.73) | 2.90 (0.70) | 2.91 (0.71)

OUTCOME MEASURES:

1. Primary Outcome: Weight Change
Description: Weight change in kilograms
Time Frame: Baseline to Post-Intervention (on average, 16 weeks)
Population: Of those who initiated the intervention, 40 individuals completed all 8 sessions and had weight data at session 8.
Measure: Mean (95% Confidence Interval); unit: kilograms
Arm/Group | Standard Care | ACT Intervention
Number analyzed (Participants) | 21 | 19
kilograms | 1.56 [-7.49 to 10.62] | 0.71 [-2.32 to 3.76]

2. Primary Outcome: Emotional Eating Change
Description: Assessed by the Dutch Eating Behavior Questionnaire (DEBQ) emotional eating subscale. Scores range from 1 (never) to 5 (very often). Lower scores reflect lower emotional eating. This subscale score is calculated by taking the mean of all items on the subscale. Negative change scores reflect decreases in emotional eating.
Time Frame: Baseline to Post-Intervention (on average, 16 weeks)
Population: Of those who initiated the intervention, only 26 participants completed the DEBQ at baseline and post-intervention (session 8) to be included in the analyses.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Standard Care | ACT Intervention
Number analyzed (Participants) | 13 | 13
units on a scale | -0.92 [-1.35 to -0.49] | -0.91 [-1.47 to -0.35]

3. Secondary Outcome: Body Fat Percentage Change
Description: Change in body fat percentage
Time Frame: Baseline to Post-Intervention (on average, 16 weeks)
Population: Of those who initiated the intervention, 40 individuals completed all 8 sessions and had body fat data at session 8.
Measure: Mean (95% Confidence Interval); unit: percentage of body fat
Arm/Group | Standard Care | ACT Intervention
Number analyzed (Participants) | 21 | 19
percentage of body fat | -0.72 [-1.53 to 0.09] | 0.16 [-0.92 to 1.23]

4. Secondary Outcome: External Eating Change
Description: Assessed by the Dutch Eating Behavior Questionnaire (DEBQ) external eating subscale. Scores range from 1 (never) to 5 (very often). Lower scores reflect lower external eating. This subscale score is calculated by taking the mean of all items on the subscale. Negative change scores reflect decreases in external eating.
Time Frame: Baseline to Post-Intervention (on average, 16 weeks)
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Standard Care | ACT Intervention
Number analyzed (Participants) | 13 | 13
units on a scale | -0.52 [-0.98 to -0.06] | -0.31 [-0.78 to 0.16]

5. Secondary Outcome: Restraint Eating Change
Description: Assessed by the Dutch Eating Behavior Questionnaire (DEBQ) restraint eating subscale. Scores range from 1 (never) to 5 (very often). Lower scores reflect lower restraint eating. This subscale score is calculated by taking the mean of all items on the subscale. Positive change scores reflect increase in restraint eating.
Time Frame: Baseline to Post-Intervention (on average, 16 weeks)
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Standard Care | ACT Intervention
Number analyzed (Participants) | 13 | 13
units on a scale | 0.27 [-0.01 to 0.55] | 0.26 [-0.16 to 0.68]

6. Secondary Outcome: Distress Tolerance Change
Description: Assessed by the Distress Tolerance Scale (DTS). All items were rated on a 5-point Likert scale from 1 (strongly agree) to 5 (strongly disagree). The score is calculated as the mean of all items. Higher scores reflect higher levels of distress tolerance. Positive change scores reflect increases in distress tolerance.
Time Frame: Baseline to Post-Intervention (on average, 16 weeks)
Population: Of those who initiated the intervention, only 26 participants completed the DTS at baseline and post-intervention (session 8) to be included in the analyses.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Standard Care | ACT Intervention
Number analyzed (Participants) | 13 | 13
units on a scale | 0.52 [0.18 to 0.86] | 0.04 [-0.31 to 0.39]

7. Secondary Outcome: Mindfulness Awareness Change
Description: Assessed by the Philadelphia Mindfulness Scale (PHLMS). All items were rated on a 5-point Likert scale from 1 (never) to 5 (very often). The subscale score is calculated as the sum of all items on the subscale, with the minimum possible score being 10 and the maximum possible score being 50. Higher scores reflect higher levels of awareness. Negative change scores reflect decreases in mindfulness and positive change scores reflect increases in mindfulness.
Time Frame: Baseline to Post-Intervention (on average, 16 weeks)
Population: Of those who initiated the intervention, only 26 participants completed the PHLMS at baseline and post-intervention (session 8) to be included in the analyses.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Standard Care | ACT Intervention
Number analyzed (Participants) | 13 | 13
units on a scale | -1.50 [-4.51 to 1.51] | 1.67 [-1.76 to 5.10]

8. Secondary Outcome: Values Clarification/ACT Application Change
Description: This questionnaire was developed for the present study to evaluate participants' real world application of the intervention. Participants were asked to indicate their level of agreement on a 5-point scale (1 = strongly agree and 5 = strongly disagree) to prompts such as "My values motivate me to lose weight" and "I am able to accept negative emotions and don't have to eat when I'm feeling bad". Total score was calculated as the mean of all items. Lower scores indicate higher values clarification. Negative change scores reflect increases in ACT application and values clarification.
Time Frame: Baseline to Post-Intervention (on average, 16 weeks)
Population: Of those who initiated the intervention, only 26 participants completed the ACT application at baseline and post-intervention (session 8) to be included in the analyses.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Standard Care | ACT Intervention
Number analyzed (Participants) | 13 | 13
units on a scale | -0.60 [-1.15 to -0.04] | -0.43 [-1.06 to 0.20]

9. Other Pre Specified Outcome: Patient Treatment Satisfaction
Description: Assessed by a self-developed questionnaire with items such as "the program reduced my emotional eating" and "the program was easy to follow". Scores represent mean ratings on a 5-point Likert-type rating scale from 1 (strongly agree) to 5 (strongly disagree). Lower scores reflect higher treatment satisfaction.
Time Frame: Administered Post-Intervention (at on average, 16 weeks)
Population: Of those who initiated the intervention, only 28 participants completed the treatment satisfaction questionnaire at post-intervention (session 8) to be included in the analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Care | ACT Intervention
Number analyzed (Participants) | 15 | 13
units on a scale | 1.95 (0.80) | 2.03 (0.77)

10. Other Pre Specified Outcome: Physician Treatment Satisfaction
Description: Assessed by a self-developed questionnaire with items such as "ease of difficulty" and "required preparation time". The following questions were assessed on Likert scales from 1 (to little) to 5 (too much) with middle scores (3) reflecting perceived balance (e.g., not too difficult, the right amount of preparation time). Total score was calculated as the mean of all items.
Time Frame: Each physician was asked to complete this questionnaire once during their administration of the ACT intervention (from July 2016 to February 2017)
Population: Physicians who delivered the ACT intervention were asked to provide their input on the intervention. They only completed this questionnaire in relation to the ACT intervention and not standard care.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- ACT Intervention: Physician treatment satisfaction for the ACT intervention.
Arm/Group | ACT Intervention
Number analyzed (Participants) | 7
units on a scale | 3.51 (0.76)

11. Other Pre Specified Outcome: Recruitment Rates
Description: Percentage of individuals who were eligible to participate in the study (based on the initial prescreen) that actually enrolled.
Time Frame: Prescreen questionnaire to Baseline
Population: 123 of those who completed the initial prescreen questionnaire were deemed eligible for the study and randomized to standard care (64) or ACT intervention (59). Of these, 43 and 44 participants, respectively actually began the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | ACT Intervention
Number analyzed (Participants) | 64 | 59
Participants | 43 | 44

12. Other Pre Specified Outcome: Number of Participants That Dropped Out From Study
Description: Dropout rates between conditions from baseline to session 8.
Time Frame: Baseline to Post-Intervention (on average, 16 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | ACT Intervention
Number analyzed (Participants) | 43 | 44
Participants | 22 | 25

13. Other Pre Specified Outcome: Questionnaire Completion
Description: Percentage of participants who completed questionnaires between conditions
Time Frame: Baseline to Post-Intervention (on average, 16 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | ACT Intervention
Number analyzed (Participants) | 43 | 44
Participants | 15 | 13

14. Other Pre Specified Outcome: Intervention Completion Time
Description: How long it took participants in each condition to complete the 8-session intervention
Time Frame: Baseline to Post-Intervention (on average, 16 weeks)
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Standard Care | ACT Intervention
Number analyzed (Participants) | 21 | 19
weeks | 15.41 (10.97) | 17.41 (12.39)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the duration which each participant was assessed, from Baseline to Post-Intervention (on average, 16 weeks).
Arm/Group | Standard Care | ACT Intervention
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/44
Other Adverse Events (participants affected / at risk) | 0/43 | 0/44

LIMITATIONS AND CAVEATS:
The intervention was terminated due to low recruitment, high attrition, and potential lack of treatment fidelity on the part of the intervening physicians.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-13): https://cdn.clinicaltrials.gov/large-docs/29/NCT03611829/Prot_SAP_002.pdf